CLINICAL TRIAL: NCT06926257
Title: Effects of VR-based Respiratory Training on Motor Reaction Time and Correctness, Stress Levels, Attention, Motor Skills, Postural Stability and Sleep Quality in Shift Healthcare Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 165/25
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Healthcare Workers; Stress Level; Emergency Department; Shift Work Sleep Disorder; Postural Stability; VR Breathing Exercises; Attention; Time Reaction
MeSH Terms: conditions — Emergencies; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (A) - no intervention (No Intervention): All participants will first be measured before and after their first night's duty to determine the baseline level of the accepted variables. Subsequently, the subjects will be informed not to use any additional forms of relaxation, and after four weeks, the study participants will undergo a final measurement.
- Experimental group (B) - breathing training using VR (Experimental): Breathing training in the experimental group will be carried out under controlled conditions, in a quiet room, using VR goggles and the Flowborne VR - Biofeedback Breathing Meditation application. The goal of the program is to learn conscious breathing and reduce stress levels through an immersive virtual reality environment.
  * A total of 8 sessions over 4 weeks.
  * 2 trainings per week (after the end of night duty).
  * Each session lasts 20 minutes.
  Interventions: Other: Experimental group (C) - breathing training using relaxation music
- Experimental group (C) - breathing training using relaxation music (Experimental): Breathing training will be based on traditional relaxation methods using relaxation music. This program will be conducted under controlled conditions in a quiet room, without the use of VR technology.
  * A total of 8 sessions over 4 weeks.
  * 2 trainings per week (after the end of night duty).
  * Each session lasts 20 minutes.
  Interventions: Other: Experimental group (B) - breathing training using VR

INTERVENTIONS:
Other: Experimental group (B) - breathing training using VR — The Flowborne VR - Biofeedback Breathing Meditation game is an interactive training environment that guides the participant through a series of breathing exercises. The app adjusts the difficulty level and pace of the workout in real time based on the participant's physiological parameters, such as breathing rhythm.
  Types of exercises in the game:
  1. diaphragmatic breathing - the participant takes slow, controlled breaths, inhaling into the diaphragm and exhaling at a set pace. The game visualizes breathing through animations of water waves and background color changes.
  2. rhythmic breathing - the participant sts his breathing rhythm to the changing visual and audio stimuli, allowing for synchronous breathing control.
  3. Controlled exhalation lengthening - the participant learns the technique of slow exhalation of air to improve relaxation and reduce tension.
  Arms: Experimental group (C) - breathing training using relaxation music
Other: Experimental group (C) - breathing training using relaxation music — * Diaphragmatic breathing - the conscious engagement of the diaphragm in the inhalation process.
  * Controlled exhalation lengthening - a technique to lengthen the exhalation phase.
  * Rhythmic breathing - synchronizing breathing with a set pace to improve breath control.
  Structure of each session:
  1. introductory phase (3 minutes)
     * Participants assume a comfortable sitting or lying position.
     * Brief instruction on proper breathing.
  2. training phase (15 minutes).
     * Participants listen to relaxation music while focusing on the breathing techniques they learned before the session.
     * Breathing techniques used include those learned during the training: diaphragmatic breathing, controlled expiration lengthening, rhythmic breathing.
       3 Relaxation phase (2 minutes)
     * Gradual exit from the training session, focusing attention on the sensations of the body and mind.
  Arms: Experimental group (B) - breathing training using VR

SUMMARY:
This study investigates the effects of virtual reality (VR)-based respiratory training on various physiological and cognitive functions in shift-working healthcare professionals, including paramedics and nurses. The research will evaluate how VR-guided breathing exercises influence: stress levels, motor reaction time and accuracy, attention and cognitive performance, motor skills and postural stability, sleep quality

Participants will be divided into three groups:

VR-based respiratory training group - performing guided breathing exercises in a VR environment.

Music-based relaxation group - listening to relaxing music without structured breathing instructions.

Control group - no intervention.

The findings will help determine whether VR-based respiratory training is an effective method for improving stress resilience, cognitive function, and physical performance in shift-working healthcare professionals.

ELIGIBILITY:
The study will be conducted in a group of paramedics and nurses of both sexes, aged 23-45. It is expected that 60 people will be examined. The study will include hospital emergency department employees, working shifts, with a minimum of two years of work experience. Those who receive a doctor's consent to participate in the study and give informed consent will be admitted to the study.

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Attention and reaction time | At the beginning of the study and after 4 weeks of breathing exercises.
  he MOXO Test is a computer-based diagnostic tool used to assess attention and impulse control. Participants respond to various visual and auditory stimuli appearing on the screen, where they must quickly and accurately recognize those that require a response while ignoring others designed to distract them. The test lasts approximately 15-18 minutes and evaluates four key indicators: reaction time, impulsivity, hyperactivity, and inattention. This allows for a detailed analysis of the participant's cognitive abilities and identification of potential attention deficits.
Postural stability | At the beginning of the study and after 4 weeks of breathing exercises.
  The assessment will be conducted using a standard, low, stable posturographic platform. The first measurement will be taken in an upright posture with an attempt to lean the body as far forward and backward as possible while maintaining stability. The second measurement involves standing on one leg.
Sleep quality | At the beginning of the study and after 4 weeks of breathing exercises.
  The impact of the intervention on participants' sleep quality, particularly in the context of shift work, will be assessed using the Polish version of the Pittsburgh Sleep Quality Index (PSQI). This measurement will be conducted twice: before the first night shift and before the last night shift (Mollayeva et al., 2016).
Stress level and mood | At the beginning of the study and after 4 weeks of breathing exercises.
  Stress levels will be assessed using the PSS-10 Perceived Stress Scale (Cohen S., Kamarck T., Mermelstein R., 1983), adapted to Polish (Juczyński Z., Ogińska-Bulik N., 2009), which evaluates the intensity of stress related to one's life situation over the past month (Matuszczak-Świgoń et al., 2023). Additionally, the PANAS (Positive and Negative Affect Schedule) questionnaire will be used to measure participants' positive and negative affect, assessing the intensity of their emotions before and after the intervention (Piotr Brzozowski, 2019). Subjective mood and the intensity of its changes will also be evaluated using a 0-10 scale before each measurement.
Fine motor skills precision | At the beginning of the study and after 4 weeks of breathing exercises.
  Fine motor skills precision will be assessed using the WorkAbility Rate of Manipulation Test (WRMT). This test is a tool for evaluating manual skills in a work-related context. It consists of a task requiring participants to transfer discs from one place to another, measuring precision, speed, and dexterity. WRMT is used in the assessment of manual task performance abilities in various industries, including vocational rehabilitation and work capacity evaluation (Wang et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The decision on data sharing has not been finalized. The availability of individual participant data (IPD) and supporting documents will be assessed after the study is completed. If data sharing is approved, details regarding access, format, and conditions will be provided in future updates.